CLINICAL TRIAL: NCT05068804
Title: Intermittent Cooling During Baseball Games Alleviated Perceived Exertion But Had no Effect on Hitting and Defense Performance in Hot Environment
Brief Title: Intermittent Cooling During Baseball Games on Hitting and Defense Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Chen Kang, Professor, National Taiwan Sport University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 18-076-A
Record Dates: First submitted 2021-09-06; First posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Decline, Cognitive
Keywords: baseball; cognitive; cooling
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cool-Down Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cooling (Experimental): The participants in the cooling trial put cold towels on their forehead and neck for 3 min in the shaded dugout during their offensive half innings when they were not scheduled to hit or on base. Each participant received the cooling intervention 3 to 4 times in each game. After each use, the towels were kept in a cooler that contained water mixed with ice and salt to keep the temperature at approximately 0℃.
  Interventions: Procedure: Cooling
- Control (Placebo Comparator): The participants in the control trial sat in the shaded dugout without any cooling intervention.
  Interventions: Other: control

INTERVENTIONS:
Procedure: Cooling — The participants in the cooling trial put cold towels on their forehead and neck for 3 min in the shaded dugout during their offensive half innings when they were not scheduled to hit or on base. Each participant received the cooling intervention 3 to 4 times in each game. After each use, the towels were kept in a cooler that contained water mixed with ice and salt to keep the temperature at approximately 0℃.
  Arms: cooling
Other: control — The participants in the control trial sat in the shaded dugout without any cooling intervention.
  Arms: Control

SUMMARY:
This study adopted a practical approach in intermittent cooling on forehead and neck during an intra-squad baseball game. Exit velocity of batted balls was used as an indicator for hitting performance and a baseball-specific reactive agility test to evaluate the cognitive performance in defense.

DETAILED DESCRIPTION:
This study used a randomized cross-over design. Each participant completed a cooling and a non-cooling trial in a random order, separated by a 20-day washout period. Each trial contained a 7-inning intra-squad game in hot environment. Hitting, reactive agility, and cognitive tests were administered before and after the game. Forehead skin and tympanic temperature, perceived exertion, and thermal sensation were measured during the game.

Experimental procedure After body weight and rectal temperature were measured in a temperature-controlled room, the participants consumed a standardized breakfast. The breakfast included white bread 1.2 g/kg, jam 0.1 g/kg, butter 0.l g/kg, and soybean milk 5 ml/kg (6.2 kcal/kg, containing carbohydrate 1.0 g/kg, protein 0.24 g/kg, and fat 0.14 g/kg). Go/NoGo and Stroop Color-Word tasks were administered after breakfast. After finishing the cognitive tests, the participants moved to the field for self-selected warm up, followed by hitting and reactive agility tests. After the intra-squad game, the participants repeated the hitting, reactive agility, and cognitive tests. The participants can drink water ad libitum during the experimental period.

Intra-squad game The 7-inning intra-squad games were played under the standard rules of baseball in hot environmental conditions (temperature 31.1-33.4℃, humidity 63-67%).

Cooling intervention The participants in the cooling trial put cold towels on their forehead and neck for 3 min in the shaded dugout during their offensive half innings when they were not scheduled to hit or on base. Each participant received the cooling intervention 3 to 4 times in each game. After each use, the towels were kept in a cooler that contained water mixed with ice and salt to keep the temperature at approximately 0℃. The participants in the control trial sat in the shaded dugout without any cooling intervention.

Measurement of temperature Rectal temperature was measured before breakfast and after the game with a digital thermometer fitted with disposable sheaths. Forehead skin and tympanic temperature were measured with infrared thermometers during their offensive half innings in the dugout.

Hitting test The participants used their own bat to hit balls thrown by a pitching machine positioned 12 m from the home plate. The ball speed was approximately 120 km/h. The participants were asked to make the best effort to hit the balls. Each test was consisted of 15 batted balls. Exit velocity was measured with a video system and swing power was measured with a sensor attached to the knob of the bat.

Reactive agility test The infielders played defense against ground balls at the short stop position while the outfielders played defense against fly balls in center field. The participants were asked to move toward the ball as soon as they determine the trajectory and make the best effort to catch it. Each test was consisted of 15 batted balls. The reaction time, the time from bat-ball contact to the participant's first definitive movement in the intended direction, was calculated post-hoc using frame-by-frame analysis of the video footage by an experienced coach

Cognitive tests The Go/NoGo and Stroop Color-Word tasks were administered on a laptop computer in a quiet room. Each task contained 100 trials.

Perceived exertion and thermal sensation The participants reported their perceived exertion and thermal sensation during their offensive half innings. Perceived exertion was estimated with a 10-point Borg scale. Thermal sensation was estimated with a 7-point scale from -3 being the coolest to 3 being the hottest.

ELIGIBILITY:
Inclusion Criteria:

* baseball players from National Taiwan University of Sport, Taiwan
* at least 6 years of experience in baseball training
* have competed nationally.

Exclusion Criteria:

* having cardiovascular or other known chronic diseases
* taking any medication in the preceding 2 months
* having musculoskeletal injuries in the preceding 2 months.

Ages: 20 Years to 23 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
rectal temperature | baseline
change in rectal temperature | 5 hours after the baseline
forehead skin temperature | baseline
change in forehead skin temperature | 2 hours after the baseline
  measured after each inning in an 2-hour 7-inning intra-squad baseball game
tympanic temperature | baseline
change in tympanic temperature | 2 hours after the baseline
  measured after each inning in an 2-hour 7-inning intra-squad baseball game
exit velocity of batted balls | baseline
change in exit velocity of batted balls | 3 hours after baseline
reactive agility in defense | baseline
  The reaction time, the time from bat-ball contact to the participant's first definitive movement in the intended direction
change in reactive agility in defense | 3 hours after baseline
  The reaction time, the time from bat-ball contact to the participant's first definitive movement in the intended direction
swing power | baseline
  power of bat swings
change in swing power | 3 hours after baseline
  power of bat swings

SECONDARY OUTCOMES:
ratings of perceived exertion | baseline
change in ratings of perceived exertion | 2 hours after baseline
  measured after each inning in an 2-hour 7-inning intra-squad baseball game
thermal sensation | baseline
change in thermal sensation | 2 hours after baseline
  measured after each inning in an 2-hour 7-inning intra-squad baseball game
Go/NoGo tasks | baseline
  reaction time and error rate
change in Go/NoGo tasks | 5 hours after baseline
  reaction time and error rate
Stroop Color-Word test | baseline
  reaction time and error rate
change in Stroop Color-Word test | 5 hours after baseline
  reaction time and error rate

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Kang Chang, Principal Investigator — National Taiwan University of Sport
Locations (1):
- National Taiwan University of Sport, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No